CLINICAL TRIAL: NCT00690703
Title: Radiofrequency Ablation of Pulmonary Tumors Response Evaluation: a Prospective, Intention-to-Treat, Multicenter Clinical Trial
Brief Title: Radiofrequency Ablation of Pulmonary Tumors Response Evaluation
Acronym: RAPTURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Riccardo Lencioni, University of Pisa, Pisa, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102-00
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Non Small Cell Lung Cancer; Pulmonary Metastases
Keywords: non small cell lung cancer; pulmonary metastases; radiofrequency ablation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment
  Interventions: Device: RF ablation (Rita Medical Systems Model 1500x)

INTERVENTIONS:
Device: RF ablation (Rita Medical Systems Model 1500x) — computed tomography-guided RF ablation with an expandable electrode needle
  Other Names: Rita Medical Systems Model 1500x; Rita Medical Systems Starburst XL

SUMMARY:
The study hypothesis is that the radiofrequency (RF) ablation is a safe and effective treatment for malignant lung tumors.

DETAILED DESCRIPTION:
Image-guided RF ablation is accepted as a viable therapeutic choice for patients with early-stage hepatocellular carcinoma or limited hepatic metastatic disease from colorectal cancer, when surgery is precluded (1, 2). Recently, RF ablation has been proposed as a viable option for the treatment of pulmonary malignancies. Experimental studies in animal tumor models have confirmed the effectiveness of RF ablation in the destruction of experimentally-induced pulmonary malignancies (3). Pilot clinical investigations have suggested that the treatment can achieve high proportions of tumor response (4, 5). We designed a prospective, intention-to-treat, multicenter clinical trial aimed at assessing feasibility, safety and effectiveness of RF ablation in the treatment of lung malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. adult (> 18 years) male or female patient
2. patient has biopsy-proven NSCLC or lung metastasis
3. patient has been rejected for surgery and has been considered unfit for radiation therapy or chemotherapy
4. patient has as many as 3 tumors per lung, each 3.5 cm or smaller in greatest diameter, by CT scan
5. tumors are located at least 1 cm from trachea; main bronchi; esophagus; aorta; aortic arch branches; pulmonary artery; and heart
6. tumors are accessible by percutaneous route
7. patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
8. patient has platelet count > 100 x 109 /L and international normalized ratio ≤ 1.5
9. patient has signed written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. patient has undergone previous pneumonectomy
2. patient is considered at high-risk for RF ablation due to major co-morbid medical conditions
3. patient has more than 3 tumors / lung
4. patient has at least one tumor > 3.5 in greatest diameter
5. tumor is associated with atelectasis or obstructive pneumonitis
6. patient has renal failure requiring hemodialysis or peritoneal dialysis
7. patient has active clinically serious infection
8. patient has history of organ allograft
9. patient has history of substance abuse or any medical, psychological or social conditions that may interfere with his / her participation in the study or evaluation of the study results
10. patient is pregnant or breast-feeding
11. patient has ECOG performance status > 2
12. patient has platelet count ≤ 100 x 109 /L or international normalized ratio > 1.5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2001-07; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
technical success | immediate
complications | 30 days
pulmonary function | 2 years
tumor response | 1 years

SECONDARY OUTCOMES:
overall survival | 2 years
cancer-specific survival | 2 years
quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Lencioni, MD, Principal Investigator — University of Pisa, Pisa, Italy
Locations (7):
- UCLA Medical Center, Los Angeles, California, United States
- University of New South Wales, Sydney, Australia
- Germany (2):
  - University Hospital Essen, Essen
  - Ludwig-Maximilians University, München
- Italy (2):
  - Institute for Cancer Research and Treatment, Candiolo
  - University of Pisa, Pisa
- University College Hospital, London, United Kingdom

REFERENCES:
- [Background] Lencioni R, Cioni D, Crocetti L, Franchini C, Pina CD, Lera J, Bartolozzi C. Early-stage hepatocellular carcinoma in patients with cirrhosis: long-term results of percutaneous image-guided radiofrequency ablation. Radiology. 2005 Mar;234(3):961-7. doi: 10.1148/radiol.2343040350. Epub 2005 Jan 21. PMID 15665226
- [Background] Tateishi R, Shiina S, Teratani T, Obi S, Sato S, Koike Y, Fujishima T, Yoshida H, Kawabe T, Omata M. Percutaneous radiofrequency ablation for hepatocellular carcinoma. An analysis of 1000 cases. Cancer. 2005 Mar 15;103(6):1201-9. doi: 10.1002/cncr.20892. PMID 15690326
- [Background] Miao Y, Ni Y, Bosmans H, Yu J, Vaninbroukx J, Dymarkowski S, Zhang H, Marchal G. Radiofrequency ablation for eradication of pulmonary tumor in rabbits. J Surg Res. 2001 Aug;99(2):265-71. doi: 10.1006/jsre.2001.6208. PMID 11469896
- [Background] Pennathur A, Luketich JD, Abbas G, Chen M, Fernando HC, Gooding WE, Schuchert MJ, Gilbert S, Christie NA, Landreneau RJ. Radiofrequency ablation for the treatment of stage I non-small cell lung cancer in high-risk patients. J Thorac Cardiovasc Surg. 2007 Oct;134(4):857-64. doi: 10.1016/j.jtcvs.2007.04.060. Epub 2007 Aug 29. PMID 17903496
- [Background] Simon CJ, Dupuy DE, DiPetrillo TA, Safran HP, Grieco CA, Ng T, Mayo-Smith WW. Pulmonary radiofrequency ablation: long-term safety and efficacy in 153 patients. Radiology. 2007 Apr;243(1):268-75. doi: 10.1148/radiol.2431060088. PMID 17392258
- [Derived] Lencioni R, Crocetti L, Cioni R, Suh R, Glenn D, Regge D, Helmberger T, Gillams AR, Frilling A, Ambrogi M, Bartolozzi C, Mussi A. Response to radiofrequency ablation of pulmonary tumours: a prospective, intention-to-treat, multicentre clinical trial (the RAPTURE study). Lancet Oncol. 2008 Jul;9(7):621-8. doi: 10.1016/S1470-2045(08)70155-4. Epub 2008 Jun 17. PMID 18565793